CLINICAL TRIAL: NCT05295576
Title: Effect of Non Surgical Periodontal Therapy on Levels of Il-17 and Il-18 in Chronic Periodontitis Patients Versus Periodontally Healthy Individuals
Brief Title: Effect of Non Surgical Periodontal Therapy on Inflammatory Markers in Chronic Periodontitis Patients
Status: Completed | Type: Observational
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Sarah Elkot, Lecturer of Oral Medicine, Periodontology and Diagnosis, Faculty of Oral and Dental Medicine, Future University in Egypt, Cairo, Egypt., Future University in Egypt
Other Study IDs: FUE12
Record Dates: First submitted 2022-03-06; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Aggressive Periodontitis
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — GCF samples collected by periopaper strips
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic periodontitis: scaling and root planing
  Interventions: Procedure: non surgical periodontal therapy
- Periodontally healthy individuals: no treatment

INTERVENTIONS:
Procedure: non surgical periodontal therapy — Scaling and root planing
  Groups: chronic periodontitis

SUMMARY:
The current study was performed to study levels of Il-17 and Il-18 in aggressive periodontitis patients before and after non surgical periodontal therapy

DETAILED DESCRIPTION:
Background:host defense factors are involved in pathogenesis of chronic periodontitis so, the current study is assessing levels of Il-17 and Il-18 in chronic periodontitis patients versus periodontally healthy controls.

Subjects and methods: Fifty subjects were included; twenty five of them are diagnosed with chronic periodontitis patients and twenty five are periodontally healthy subjects. Probing depth (PD), clinical attachment level (CAL), plaque index (PI) and gingival index (GI) were recorded for all the enrolled subjects. GCF levels of Il-17 and IL-18 were analyzed by enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Medically free subjects .
* both genders .
* age range between 30 to 60 years old .

Exclusion Criteria:

* Subjects with periodontal surgeries in the last 6 months.
* Subjects with prior use of antibiotics in the last 6 months.
* Smokers.
* Pregnant and lactating females were excluded.
* Lactating females.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Chronic periodontitis patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
measure levels of Il-17 and Il-18 in chronic periodontitis patients | Change from Baseline Il-17 andIl-18 at 3 months
  measure levels of Il-17 and Il-18 in GCF of chronic periodontitis patients

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Elkot, Lecturer, Principal Investigator — Lecturer of Oral Medicine and Periodontology
Locations (1):
- Future university in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided